CLINICAL TRIAL: NCT01240148
Title: A Randomised, Double-Blind, Placebo-Controlled, Single-Centre Study to Determine the Effect of Intradermal AZD3161 on Quantitative Sensory Testing Variables in Normal and UVC Exposed Skin in Healthy Volunteers
Brief Title: Determine the Effect of AZD3161,Injected Intradermally, on Quantitative Sensory Testing Variables in Normal and Ultraviolet-C (UVC) Exposed Skin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: D3780C00005
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Peripheral Neuropathic Pain; Nociceptive Pain
Keywords: Allodynia; hyperalgesia; paresthesia
MeSH Terms: conditions — Nociceptive Pain; Hyperalgesia; Paresthesia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 1 (Experimental): 150 μL intradermal injection of 1 μmol/L AZD3161
  Interventions: Drug: AZD3161
- 2 (Experimental): 150 μL intradermal injection of 6 μmol/L AZD3161
  Interventions: Drug: AZD3161
- 3 (Experimental): 150 μL intradermal injection of 30 μmol/L AZD3161
  Interventions: Drug: AZD3161
- 4 (Active Comparator): 150 μL intradermal injection of 10 mg/mL Lidocaine
  Interventions: Drug: Lidocaine
- 5 (Placebo Comparator): 150 μL intradermal injection of AZD3161 placebo
  Interventions: Drug: AZD3161 Placebo

INTERVENTIONS:
Drug: AZD3161 — Single dose, intradermal injection
  Arms: 1; 2; 3
Drug: Lidocaine — Single dose, intradermal injection
  Arms: 4
Drug: AZD3161 Placebo
  Arms: 5

SUMMARY:
The purpose of this study is to investigate the effect of AZD3161 on mechanical pain sensitivity and axon reflex flare in normal and ultraviolet C irradiated skin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian male and female volunteers aged 18 to 55 years inclusive with suitable veins for venepuncture
* The subject belongs to skin type II or III according to Fitzpatrick skin type scale
* Females must have a negative pregnancy test at screening and at admission, must not be lactating and must be of non-child-bearing potential
* Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh between 50 kg and 100 kg inclusive
* Male subjects should be willing to use barrier contraception ie, condoms, from the day of dosing until 3 months after dosing with investigational product.

Exclusion Criteria:

* Presence of skin disorders, tattoos or other skin conditions that may interfere with the QST measurements, as judged by the Investigator
* Recent exposure to significant amount of UV light, as judged by the Investigator.
* Use of any prescribed or non-prescribed analgesics (including paracetamol/acetaminophen or drugs affecting blood flow (including nasal anticongestants), prior to the first administration of investigational product that may interfere with the study objectives.
* History of severe allergy/hypersensitivity, or ongoing allergy/hypersensitivity as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to AZD3161.
* Plasma donation within 1 month of screening or any blood donation/blood loss >500 mL during the 3 months prior to screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Results of mechanical pain testing using Quantitative Sensory Testing | Day 1

SECONDARY OUTCOMES:
Number of participants with Adverse Events | Range of 14 days
Vital signs | Day 1
  (blood pressure, heart rate, pulse)
Clinical chemistry (urinalysis, hematology) | At follow up (a range of 8-15 days after Day 1)
The effect of AZD3161 on axon reflex flare in normal and UVC irradiated skin using a Laser doppler scan | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, MD, MBBS DCPSA, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital; Bo Fransson, Study Chair — AstraZeneca R&D
Locations (1):
- Research Site, London, United Kingdom